CLINICAL TRIAL: NCT01032070
Title: A Randomized, Phase 2 Study of Single-agent Erlotinib Versus Oral Etoposide in Patients With Recurrent or Refractory Pediatric Ependymoma
Brief Title: Erlotinib Versus Oral Etoposide in Patients With Recurrent or Refractory Pediatric Ependymoma
Acronym: PETEY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In a pre-planned interim analysis, OSI-774-205 met futility for efficacy with no safety concerns. As a result, it has been stopped.
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-205; 2009-016836-11 (EudraCT Number)
Record Dates: First submitted 2009-12-10; First posted 2009-12-15 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Recurrent or Refractory Pediatric Ependymoma
Keywords: pediatric; etoposide; erlotinib; phase 2; ependymoma
MeSH Terms: conditions — Recurrence; Familial ependymoma; Ependymoma | interventions — Erlotinib Hydrochloride; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib (Experimental): Erlotinib was administered orally at a dose of 85 mg/m^2 per day continuously until either progression, death, patient request or investigator decision to discontinue study drug or intolerable toxicity.
  Interventions: Drug: erlotinib
- Etoposide (Active Comparator): Etoposide 50 mg/m^2 per day was administered orally for 21 days followed by a 7-day rest period until either progression, death, patient request or investigator decision to discontinue study drug or intolerable toxicity.
  Interventions: Drug: etoposide

INTERVENTIONS:
Drug: erlotinib — oral
  Other Names: OSI-774; Tarceva
  Arms: Erlotinib
Drug: etoposide — oral
  Other Names: VP-16
  Arms: Etoposide

SUMMARY:
This is a phase 2 study to evaluate the efficacy of single-agent erlotinib versus oral etoposide in patients with recurrent or refractory pediatric ependymoma.

DETAILED DESCRIPTION:
This is a phase 2 study involving a 1:1 randomization of 40 patients with recurrent or refractory pediatric ependymoma who will receive either erlotinib or oral etoposide.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent of refractory ependymoma or subependymoma
* Performance Status (PS): Lansky ≥ 50% for patients ≤ 10 years of age or Karnofsky ≥ 50% for patients >10 years of age
* Measurable disease, defined as 1 measurable lesion that can be accurately measured in 2 planes that has not received radiation therapy within 12 weeks
* Recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* ≥ 1 year to ≤ 21 years
* Serum creatinine for patients ≤ 5 years in age is ≤ 0.8 mg/dL or Creatinine Clearance/Glomerular Filtration Rate (GFR) ≥ 70 mL/min/m^2
* Serum creatinine for patients > 5 and ≤ 10 years in age is ≤ 1.0 mg/dL or Creatinine Clearance/GFR ≥ 70 mL/min/m^2
* Serum creatinine for patients > 10 and ≤ 15 years in age is ≤ 1.2 mg/dL or Creatinine Clearance/GFR ≥ 70 mL/min/m^2
* Serum creatinine for patients > 15 years in age is ≤ 1.5 mg/dL or Creatinine Clearance/GFR ≥ 70 mL/min/m^2
* Total bilirubin is ≤ 1.5 x upper limit of normal for age
* Alanine aminotransferase (ALT) ≤ 3 x upper limit of normal
* Absolute neutrophil count > 1000/µL
* Platelet count > 100,000/µL
* Hemoglobin > 8 gm/dL
* Neurologically stable for at least 7 days prior to randomization
* If receiving corticosteroids, patients must be on a stable or decreasing dose for at least 7 days before randomization
* Patients of reproductive potential must agree to proactive effective contraceptive measures for the duration of the study and for at least 90 days after completion of study drug

Exclusion Criteria:

* Previously received epidermal growth factor receptor (EGFR)-targeted therapy
* Previously received oral etoposide
* Received craniospinal radiotherapy within 24 weeks prior to randomization
* Received field radiotherapy to the target lesion within 12 weeks prior to randomization
* Received symptomatic metastatic disease within 14 days prior to randomization
* Received myelosuppressive chemotherapy within 21 days before randomization
* Received growth factors within 7 days prior to randomization
* Participating in another investigational drug trial
* Received a biologic agent within 7 days prior to randomization
* Received a monoclonal antibody within 28 days prior to randomization
* Taking cytochrome P450 (CYP)3A4 or CYP1A2 inhibitors/inducers within 14 days prior to randomization
* Taking proton pump inhibitors within 14 days prior to randomization
* Smoking during treatment
* Pregnant or breast-feeding females

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2012-11-26 (Actual); Study Completion 2012-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (28):
- United States (18):
  - University of Alabama at Birmingham Dept. of Pediatric-Hematology/Oncology, Birmingham, Alabama
  - Center for Cancer and Blood Disorders-Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Stanford University and Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Children's National Medical Center - D.C. Center for Cancer and Blood Disorders, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University Children's Healthcare of Atlanta Aflac Cancer Center & Blood Disorders, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute Department of Pediatric Neuro-oncology, Boston, Massachusetts
  - Amplatz Children's Hospital University of Minnesota Medical Center- Pediatric Hematology Oncology, Minneapolis, Minnesota
  - Steven D Hassenfeld Children's Center - New York University, New York, New York
  - Columbia University Children's Hospital of New York Presbyterian Child & Adolescent Oncology Center, New York, New York
  - Oregon Health & Sciences University Doembecher Children's Hospital, Portland, Oregon
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center, Dallas Center for Cancer and Blood Disorders, Dallas, Texas
  - University of Wisconsin Pediatric Hematology/Oncology Department, Madison, Wisconsin
- Canada (3):
  - Strollery Children's Hospital Division of Hematology/Oncology, Edmonton, Alberta
  - Children's and Women's Health Center of BC Division of Hematology/ Oncology/ BMT, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
- United Kingdom (7):
  - Birmingham Children's Hospital, Birmingham
  - Royal Hospital for Sick Children, Glasgow
  - Paediatric Oncology and Haematology Offices, Leeds
  - Alder Hey Children's NHS Foundation Trust Department of Oncology, Liverpool
  - Royal Manchester Children's Hospital Ward 84, Manchester
  - University of Nottingham Children's Brain Tumour Research Centre, Nottingham
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=328

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib | Etoposide
Started | 13 | 12
Completed | 0 | 0
Not Completed | 13 | 12
Not completed — Disease progression | 13 | 8
Not completed — Medical or ethical reasons | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Etoposide | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (5.87) | 9.2 (4.99) | 11.1 (5.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Indian Subcontinent | 0 | 1 | 1
  Asian - Southeast Asia | 0 | 1 | 1
  Black | 1 | 1 | 2
  Other | 1 | 0 | 1
  White | 11 | 9 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 1 | 2 | 3
  Not Hispanic/Latino | 12 | 10 | 22
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.51 (0.556) | 1.17 (0.439) | 1.35 (0.521)
Tumor Type for Initial Disease Diagnosis [Number; unit: participants]
  Anaplastic Ependymoma | 6 | 9 | 15
  Ependymoma | 6 | 3 | 9
  Myxopapillary Ependymoma | 1 | 0 | 1
Total Number of Disease Recurrences [Median (Full Range); unit: recurrences] | 3 (2.1) [1 to 9] | 2 (0.8) [1 to 3] | 2 (1.7) [1 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response
Description: Objective response is defined as a best overall response of complete response (CR) or partial response (PR), evaluated using modified International Society of Pediatric Oncology Brain, Tumor Subcommittee for the Reporting of Trials criteria. Response was confirmed at least 28 days after the first assessment where the response criteria were met. Response was assessed by magnetic resonance imaging (MRI) every 8 weeks. CR: • Complete disappearance of all enhancing tumor and mass effect • On a stable or decreasing dose of corticosteroids (or receiving only adrenal replacement doses) • Stable or improving neurologic examination sustained for ≥ 4 weeks • If cerebral spinal fluid (CSF) evaluation was positive, it must become negative (confirmed at least 2 times at consecutive samplings). PR: • ≥ 50% reduction in tumor size by bi-dimensional measurement • On a stable or decreasing dose of corticosteroids • Stable or improving neurologic examination sustained for ≥ 4 weeks.
Time Frame: From randomization until the end of treatment. The median time on treatment was 52 days for erlotinib and 58 days for etoposide.
Population: The Full Analysis Set (FAS) consisted of all randomized participants. Following the intent-to-treat (ITT) principle, participants were analyzed according to the treatment arm they were assigned to at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
percentage of participants | 0 [0 to 24.7] | 16.7 [2.1 to 48.4]
Statistical Analysis 1: Comparison: Erlotinib vs Etoposide; The study was not powered for this comparison due to small sample size; Test type: Superiority or Other; p = 0.2200, Fisher Exact — P-value is not adjusted for multiple comparisons

2. Secondary Outcome: Duration of Response
Description: Duration of response (complete or partial response [CR/PR]) was defined as the time from the date of the first documented response (CR/PR) to the first documented progression or death due to underlying cancer. If a participant had not progressed or died, the duration of overall response was censored at the date of last adequate disease assessment. Duration of response was only defined for participants whose best overall response was CR or PR. Progression was defined as a worsening of neurologic status that could not be explained by other causes, a > 25% increase in tumor size, the appearance of new lesions or CSF positivity, or increasing doses of corticosteroids required to maintain stable status.
Time Frame: as for outcome 1
Population: Full Analysis Set participants whose best overall response was CR or PR.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 0 | 2
days |  | NA [NA to NA] — Two participants achieving PR were censored at 174 and 463 days, respectively.

3. Secondary Outcome: Percentage of Participants With a Minor Response
Description: Participants with a best overall response of minor response (MR), defined as: • ≥ 25% to < 50% reduction in tumor size by bi-dimensional measurement • On a stable or decreasing dose of corticosteroids • Stable or improving neurologic examination sustained for ≥ 4 weeks.
Time Frame: as for outcome 1
Population: The Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
percentage of participants | 0 [0 to 24.7] | 25.0 [5.5 to 57.2]

4. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control is a best overall response of CR or PR or MR or Stable disease (SD). CR: • Complete disappearance of all enhancing tumor and mass effect • On a stable or decreasing dose of corticosteroids • Stable or improving neurologic examination sustained for ≥ 4 weeks • If CSF evaluation was positive, it must become negative (confirmed at least 2 times consecutively). PR: • ≥ 50% reduction in tumor size by bi-dimensional measurement • On a stable or decreasing dose of corticosteroids • Stable or improving neurologic examination sustained for ≥ 4 weeks. MR: • ≥ 25% to < 50% reduction in tumor size by bi-dimensional measurement • On a stable or decreasing dose of corticosteroids • Stable or improving neurologic examination sustained for ≥ 4 weeks. SD: • Neurologic examination is at least stable • Maintenance corticosteroid dose is not increased • MRI meets neither the criteria for minor response nor for progressive disease • Sustained for ≥ 8 weeks.
Time Frame: as for outcome 1
Population: The Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
percentage of participants | 15.4 [1.9 to 45.4] | 41.7 [15.2 to 72.3]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to disease progression based on central nervous system (CNS)-specific evaluation criteria as assessed by the investigator or death due to any cause, whichever occurs first. Participants did not progress or die before the data cutoff date for analysis were censored at the date of last disease assessment (including both radiologic assessment and neurologic assessment) where non-progression was documented. If a participant received any further anticancer therapy without prior documentation of disease progression, the participant was censored at the date of last disease assessment before starting new anti-cancer treatment. Participants were also censored at the date of last disease assessment with no documented progression if patients discontinued treatment for undocumented progression, toxicity or other reason before the data cutoff date for analysis.
Time Frame: as for outcome 1
Population: The Full Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
days | 52 [29.0 to 62.0] | 65 [23.0 to NA] — Upper limit could not be estimated due to the low number of events

6. Secondary Outcome: Percentage of Participants With Prolonged Stable Disease
Description: Prolonged stable disease (SD) was defined as SD with a duration of at least 16 weeks. The percentage of participants with prolonged SD was defined as participants who achieved a best overall response of CR or PR or MR or SD, and did not progress within 16 weeks from randomization. Progression was defined as a worsening of neurologic status that could not be explained by other causes, a > 25% increase in tumor size, the appearance of new lesions or CSF positivity, or increasing doses of corticosteroids required to maintain stable status.
Time Frame: as for outcome 1
Population: The Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
percentage of participants | 0 [0 to 24.7] | 41.7 [15.2 to 72.3]

7. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease (SD; defined as participants with an overall best response of complete, partial or minor response or stable disease) was defined as the time from the date of randomization to the first documented progression or death due to underlying cancer. If a participant had not progressed or died, the duration of SD was censored at the date of last adequate disease assessment. Duration of SD was only defined for participants whose best overall response was CR or PR or MR or SD. Progression was defined as a worsening of neurologic status that could not be explained by other causes, a > 25% increase in tumor size, the appearance of new lesions or CSF positivity, or increasing doses of corticosteroids required to maintain stable status.
Time Frame: as for outcome 1
Population: Full Analysis Set participants whose best overall response was CR, PR, MR or SD.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 2 | 5
days | 79 [78 to 80] | NA [117 to NA] — Not calculable due to the low number of events (disease progression or death)

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization until the documented date of death. Participants who were still alive by the data cutoff date for analysis were censored on the last day the participant was known to be alive.
Time Frame: From randomization up to 12 months after the last dose. Median duration of follow-up was 12.9 months for erlotinib and 14.4 months for etoposide.
Population: The Full Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
days | NA [114.0 to NA] — Could not be estimated due to the low number of events. | 261 [154.0 to NA] — Could not be estimated due to the low number of events.

9. Secondary Outcome: Safety Assessed Through Evaluation of Physical Exams, Vital Signs, Clinical Laboratory Tests and Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a study participant and did not necessarily have a causal relationship with study treatment. Clinically significant vital sign assessments, findings on physical or neurological examination, and laboratory findings associated with signs and/or symptoms requiring withdrawal, dose modification or medical intervention were recorded as AEs. An AE was considered serious if it resulted in death, a life-threatening situation, inpatient hospitalization or prolongation of an existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect in the offspring of a patient who received study drug or other important medical events. The relationship of each AE to study drug was assessed as either related or not related.
Time Frame: From the date of first dose of study drug until 30 days after the last dose. The median time on treatment was 52 days for erlotinib and 58 days for etoposide.
Population: All enrolled participants who received at least 1 dose of study drug (Safety Analysis Set).
Measure: Number; unit: participants
Arm/Group | Erlotinib | Etoposide
Number analyzed (Participants) | 13 | 12
participants
  Any adverse event | 13 | 11
  Drug-related adverse event | 11 | 10
  Adverse event leading to death | 1 | 0
  Drug-related adverse event leading to death | 0 | 0
  Serious adverse event | 6 | 5
  Drug-related serious adverse event | 0 | 1
  AE leading to discontinuation | 0 | 0
  Drug-related AE leading to discontinuation | 0 | 0
  AE leading to dose interruption | 2 | 5
  Drug-related AE leading to dose interruption | 1 | 3
  AE leading to dose interruption and reduction | 1 | 2
  Related AE leading to dose interruption/ reduction | 1 | 2

10. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours Post-dose for Erlotinib
Description: Pharmacokinetic parameters were determined from the serial plasma concentration data obtained for erlotinib. Area under the plasma concentration-time curve from time zero to 24 hours (the dosing interval) measured at steady state using sparse sampling.
Time Frame: Day 14 predose and 0.5 to 1.5 hours, 2 to 3 hours and 4 to 8 hours post-dose.
Population: The Pharmacokinetics Analysis Set (PKAS) consisted of the participants treated with erlotinib for whom sufficient analyte concentration data were available to facilitate derivation of at least 1 primary pharmacokinetic parameter. Participants may have been excluded from the PKAS for reasons such as missing data or protocol deviation.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
h*ng/mL | 26716.7 [20269 to 35215.4]

11. Secondary Outcome: Maximum Observed Plasma Concentration of Erlotinib (Cmax)
Description: Pharmacokinetic parameters were determined from the serial plasma concentration data obtained for erlotinib. Maximum observed plasma concentration of erlotinib (Cmax) was measured at steady state on Day 14 using sparse sampling.
Time Frame: Day 14 predose and 0.5 to 1.5 hours, 2 to 3 hours and 4 to 8 hours post-dose.
Population: The Pharmacokinetics Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
ng/mL | 1969.5 [1627.7 to 2382.9]

12. Secondary Outcome: Time to Maximum Observed Plasma Concentration of Erlotinib (Tmax)
Description: Pharmacokinetic parameters were determined from the serial plasma concentration data obtained for erlotinib. Time to the maximum observed plasma concentration of erlotinib (Tmax) was measured at steady state on Day 14 using sparse sampling.
Time Frame: Day 14 predose and 0.5 to 1.5 hours, 2 to 3 hours and 4 to 8 hours post-dose.
Population: The Pharmacokinetics Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
hours | 2.100 [1.6 to 2.7]

13. Secondary Outcome: Apparent Body Clearance (CL/F) of Erlotinib
Description: Pharmacokinetic parameters were determined from the serial plasma concentration data obtained for erlotinib. Apparent body clearance (CL/F) of erlotinib was measured at steady state on Day 14 using sparse sampling.
Time Frame: Day 14 predose and 0.5 to 1.5 hours, 2 to 3 hours and 4 to 8 hours post-dose.
Population: The Pharmacokinetics Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/m^2
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
mL/h/m^2 | 2922.1 [2233.4 to 3823.3]

14. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Erlotinib
Description: Pharmacokinetic parameters were determined from the serial plasma concentration data obtained for erlotinib. The apparent volume of distribution (Vz/F) of erlotinib was measured at steady state on Day 14 using sparse sampling.
Time Frame: Day 14 predose and 0.5 to 1.5 hours, 2 to 3 hours and 4 to 8 hours post-dose.
Population: The Pharmacokinetics Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: mL/m^2
Arm/Group | Erlotinib
Number analyzed (Participants) | 11
mL/m^2 | 71628.5 [59572 to 86124.9]

ADVERSE EVENTS:
Time Frame: From the date of first dose of study drug until 30 days after the last dose. The median time on treatment was 52 days for erlotinib and 58 days for etoposide.
Arm/Group | Erlotinib | Etoposide
Serious Adverse Events (participants affected / at risk) | 6/13 | 5/12
Other Adverse Events (participants affected / at risk) | 13/13 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=13) | Etoposide (N=12)
Convulsion (Nervous system disorders) | 2 | 1
Hydrocephalus (Nervous system disorders) | 2 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=13) | Etoposide (N=12)
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 6 | 8
Constipation (Gastrointestinal disorders) | 3 | 6
Nausea (Gastrointestinal disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaethesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 7
Nystagmus (Nervous system disorders) | 3 | 2
Ataxia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Facial palsy (Nervous system disorders) | 1 | 1
Hypoaethesia (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Meningism (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Ageusia (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 1
Tongue paralysis (Nervous system disorders) | 0 | 1
Upper motor neurone lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 3 | 8
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 4
Mucosal inflammation (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Irritability (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Weight decreased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Optic nerve disorder (Eye disorders) | 0 | 1
Strabismus (Eye disorders) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1
Corneal infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3
urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Anthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Catheter site pain (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Epistaxis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Multiple allergies (Immune system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1
Enuresis (Renal and urinary disorders) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 2
Breast enlargement (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.